CLINICAL TRIAL: NCT05364697
Title: IonMAN Trial-First in Human Study of the IoNIR Ridaforolimus-Eluting Coronary Stent System
Brief Title: IonMAN Trial- First in Human Study of the IoNIR Ridaforolimus-Eluting Coronary Stent System
Acronym: IonMAN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medinol Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IoNIR-001
Record Dates: First submitted 2022-05-03; First posted 2022-05-06 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Coronary Stenosis; Coronary Disease; Non-ST Elevated Myocardial Infarction; Cardiovascular Diseases
MeSH Terms: conditions — Coronary Stenosis; Coronary Disease; Non-ST Elevated Myocardial Infarction; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IoNIR Ridaforolimus-Eluting Coronary Stent (Experimental): IoNIR Ridaforolimus-Eluting Coronary Stent System
  Interventions: Device: IoNIR Ridaforolimus-Eluting Coronary Stent System

INTERVENTIONS:
Device: IoNIR Ridaforolimus-Eluting Coronary Stent System — The IoNIR Ridaforolimus-Eluting Coronary Stent System is a sterile single-use device/drug combination product, comprised of a cobalt chromium (CoCr) alloy-based stent coated with a bioresorbable polymer mesh which is embedded with drug, mounted on a Rapid Exchange (RX) delivery system.
  Other Names: IoNIR

SUMMARY:
This is a prospective, multi-center, single-arm, open-label, First in Human clinical trial to provide preliminary evidence for the safety and efficacy of the novel IoNIR stent system.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Patient with an indication for PCI including NSTEMI (biomarkers have peaked or are falling), angina (stable or unstable), silent ischemia (in absence of symptoms a visually estimated target lesion diameter stenosis of ≥70%, a positive non-invasive stress test, or FFR ≤0.80, Pd/Pa≤0.91or iFR, RFR, DFR, DPR≤0.89 must be present).
3. Non-target vessel PCIs are allowed if performed >30 days prior to index procedure.
4. Patient or legal guardian is willing and able to provide informed written consent and comply with follow-up visits and testing schedule.
5. Staged procedures are allowed as long as the IoNIR stent is implanted in the last procedure and at least 30 days have elapsed between the previous procedure and the IoNIR PCI.
6. One de novo target lesion ONLY may be treated (more than one lesion separated by less than 5 mm are considered one lesion).
7. Target lesion must be in a major native coronary artery with visually estimated diameter of ≥2.5 mm to ≤4.0 mm and lesion length of up to 28 mm, and appropriate size IoNIR stent is available

Exclusion Criteria:

1. ST Segment Elevation MI within past 30 days.
2. NSTEMI with biomarkers that have not peaked.
3. Significant valvular disease or planned valvular intervention.
4. PCI within the 30 days preceding the baseline procedure.
5. PCI in the target vessel within 12 months of the baseline procedure.
6. Planned staged procedures (coronary or valvular), where the study stent is implanted in the first stage.
7. Brachytherapy in conjunction with the baseline procedure.
8. Known history of stent thrombosis.
9. Cardiogenic shock (defined as persistent hypotension (systolic blood pressure <90 mm/Hg for more than 30 minutes) or requiring pressors or hemodynamic support, including IABP.
10. Subject is intubated.
11. Known LVEF <30%.
12. Relative or absolute contraindication to DAPT for 6 months in non-ACS patients and 12 months in ACS patients (including planned surgeries that cannot be delayed).
13. Subject has an indication such as atrial fibrillation for oral anticoagulation/prolonged heparinization (i.e., use of coumadin/DOAC (NOAC) or prolonged enoxaparin/heparin therapy is not allowed).
14. eGFR <60 mL/min.
15. Hemoglobin <10 g/dL.
16. Platelet count <100,000 cells/mm3 or >700,000 cells/mm3.
17. White blood cell (WBC) count <3,000 cells/mm3.
18. Clinically significant liver disease.
19. Active peptic ulcer or active bleeding from any site
20. Bleeding from any site within the previous 8 weeks requiring active medical or surgical attention.
21. If femoral access is planned, significant peripheral arterial disease which precludes safe insertion of a 6F sheath.
22. History of bleeding diathesis or coagulopathy and patients that refuse blood transfusions.
23. Cerebrovascular accident or transient ischemic attack within the past 6 months, or any permanent neurologic defect attributed to CVA.
24. Known allergy to the study stent components (cobalt, nickel, chromium, molybdenum, PDLG, PLC, or limus drugs (ridaforolimus, zotarolimus, tacrolimus, sirolimus, everolimus, or similar drugs or any other analogue or derivative or similar compounds).
25. Known allergy to protocol-required concomitant medications such as aspirin, or P2Y12 inhibitors (clopidogrel, prasugrel, and ticagrelor), heparin and bivalirudin, or iodinated contrast allergy that cannot be adequately pre-medicated.
26. Any co-morbid condition that may cause non-compliance with the protocol (e.g., dementia, substance abuse, etc.) or reduced life expectancy to <24 months (e.g., cancer, severe heart failure, severe lung disease).
27. Patient is participating in or plans to participate in any other investigational drug or device clinical trial that has not reached its primary endpoint.
28. Women who are pregnant or breastfeeding.
29. Women who intend to become pregnant within 12 months after the baseline procedure (women of child-bearing potential who are sexually active must agree to use a reliable method of contraception from the time of screening through 12 months after the baseline procedure).
30. Patient has received an organ transplant or is on a waiting list for an organ transplant.
31. Patient is receiving or scheduled to receive chemotherapy within 30 days before or any time after the baseline procedure.
32. Patient is receiving oral or intravenous immunosuppressive therapy or has known life-limiting immunosuppressive or autoimmune disease (e.g., HIV). Corticosteroids are allowed
33. More than one lesion of greater than 50% stenosis in the target vessel.
34. Complex lesions including severely calcified lesions, lesions requiring scoring/cutting and/or rotational/orbital atherectomy and/or intra-vascular lithotripsy, presence of visible thrombus, chronic total occlusions, bifurcation lesions (side branch diameter ≥2.0 mm), tortuous lesions, restenotic lesions, left main lesions, ectasia, aneurysm and any bypass graft lesions.
35. Another lesion in a target or non-target vessel (including all side branches) is present that requires or has a high probability of requiring PCI within 12 months after the baseline procedure.
36. Ostial lesions within 3 mm of LAD, LCx, RCA ostia, lesions in the LM

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-30 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
1In-stent Late Loss (LL) | 1 year
  In-stent Late Loss (LL) at 1 year (cohort B) assessed by quantitative coronary angiography (QCA) (Minimal Lumen Diameter (MLD) post-procedure - MLD follow-up)
Target Lesion Failure | 1 year
  Target Lesion Failure (composite of cardiovascular death, target vessel-related myocardial infarction, or ischemia-driven target lesion revascularization) at 1 year

SECONDARY OUTCOMES:
Major adverse cardiac events | 30 days, 6 months, 1, 2, 3, 4, 5 years
  Major adverse cardiac events (MACE; the composite rate of cardiovascular death, any MI or ischemia-driven target lesion revascularization (TLR))
All-cause mortality | 30 days, 6 months, 1, 2, 3, 4, 5 years
  All-cause mortality.
Cardiovascular death | 30 days, 6 months, 1, 2, 3, 4, 5 years
  Cardiovascular death.
Myocardial infarction | 30 days, 6 months, 1, 2, 3, 4, 5 years
  Myocardial infarction.
Target vessel related MI | 30 days, 6 months, 1, 2, 3, 4, 5 years
  Target vessel related MI.
Target Lesion Failure | 6 months, 2, 3, 4, 5 years
  Target Lesion Failure (TLF)
Ischemia-driven TLR | 30 days, 6 months, 1, 2, 3, 4, 5 years
  Ischemia-driven Target Lesion Revascularization
Ischemia-driven Target Vessel Revascularization | 30 days, 6 months, 1, 2, 3, 4, 5 years
  Ischemia-driven Target Vessel Revascularization.
Stent thrombosis | 30 days, 6 months, 1, 2, 3, 4, 5 years
  Stent thrombosis (ARC-2 definite and probable)
Acute Device Success | index procedure
  Acute Device Success (successful crossing and deployment with residual QCA DS <30%).
Luminal gain | Cohort A: 30 days Cohort B: 12 months
  Luminal gain (MLD post-procedure - MLD pre-procedure).
In-stent MLD | Cohort A: 30 days Cohort B: 12 months
  In-stent Minimal Lumen Diameter
In-segment MLD | Cohort A: 30 days Cohort B: 12 months
  In-segment (+5mm from the stent edges) MLD
In-segment late loss | Cohort A: 30 days Cohort B: 12 months
  In-segment (+5mm from the stent edges) late loss
Proximal late loss | Cohort A: 30 days Cohort B: 12 months
  Proximal late loss (+5 mm from proximal stent edge)
Distal late loss | Cohort A: 30 days Cohort B: 12 months
  Distal late loss (+5 mm from distal stent edge)
In-stent and in-segment Binary Restenosis | Cohort A: 30 days Cohort B: 12 months
  In-stent and in-segment Binary Restenosis.
OCT-determined inner layer percent neointimal hyperplasia volume | Cohort A: 30 days Cohort B: 12 months
  CT-determined inner layer percent neointimal hyperplasia volume.
In-stent MLA | Cohort A: 30 days Cohort B: 12 months
  In-stent Minimum Lumen Area
In-segment minimum lumen area | Cohort A: 30 days Cohort B: 12 months
  In-segment minimum lumen area (MLA)
Minimal stent area | Cohort A: 30 days Cohort B: 12 months
  Minimal stent area (MSA)
Stent expansion | Cohort A: 30 days Cohort B: 12 months
  Stent expansion.
Edge dissection | Cohort A: 30 days Cohort B: 12 months
  Edge dissection.
NIH percentage at the MLA | Cohort A: 30 days Cohort B: 12 months
  NIH (Neointimal hyperplasia) percentage at the MLA
Percentage of Area stenosis at the MLA | Cohort A: 30 days Cohort B: 12 months
  Percentage of Area stenosis at the MLA.
Luminal gain | Cohort A: 30 days Cohort B: 12 months
  Luminal gain (MLA post-procedure - MLA pre-procedure)
In-stent late loss MLA | Cohort A: 30 days Cohort B: 12 months
  In-stent late loss MLA.
In-segment (+5 mm from the stent edges) late loss (MLA) | Cohort A: 30 days Cohort B: 12 months
  In-segment (+5 mm from the stent edges) late loss (MLA).
Proximal late loss (+5 mm from proximal stent edge) (MLA) | Cohort A: 30 days Cohort B: 12 months
  Proximal late loss (+5 mm from proximal stent edge) (MLA).
Distal late loss (+5 mm from distal stent edge) (MLA) | Cohort A: 30 days Cohort B: 12 months
  Distal late loss (+5 mm from distal stent edge) (MLA).
Intraluminal mass at least 0.2 mm beyond the luminal edge of a strut | Cohort A: 30 days Cohort B: 12 months
  Intraluminal mass at least 0.2 mm beyond the luminal edge of a strut (Intraluminal mass attached to the vessel is defined as an irregularly shaped structure in contact with the luminal contour, a free intraluminal mass is defined as an isolated structure in the lumen without contact to the vessel wall)
Malapposition | Cohort A: 30 days Cohort B: 12 months
  Malapposition (stent struts clearly separated from the vessel wall (lumen border/plaque surface) without tissue behind the struts with a distance from the adjacent intima of ≥0.2 mm not associated with any side branch)
Percentage of Covered strut | Cohort A: 30 days Cohort B: 12 months
  Percentage of Covered strut (NIH thickness of >0 μm)
Percentage of Healthy covered strut | Cohort A: 30 days Cohort B: 12 months
  Percentage of Healthy covered strut (NIH thickness≥40 μm)
Peri-strut low intensity area | Cohort A: 30 days Cohort B: 12 months
  Peri-strut low intensity area (peri-strut region of homogeneous lower intensity observed without signal attenuation)
Healing score | Cohort A: 30 days Cohort B: 12 months
  Healing score (defined as % intraluminal mass [=intraluminal mass volume/stent volume] ×4 + % malposed and uncovered struts ×3 + (% uncovered struts alone ×2 + % malposed struts alone ×1)
  1. Intraluminal mass (+4).
  2. Malposed and uncovered struts (+3).
  3. Uncovered struts alone (+2).
  4. Malposed struts alone (+1)

CONTACTS AND LOCATIONS:
Locations (4):
- InCor, São Paulo, Brazil
- Israel (3):
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: Undecided